CLINICAL TRIAL: NCT06900335
Title: Characterization of the Functional Connectome in Prader-Willi Syndrome: Integrating Neuroimaging and Artificial Intelligence to Assess the Impact of Physiological and Therapeutic Interventions
Brief Title: Functional Connectome in Prader-Willi Syndrome: Neuroimaging and AI to Assess Therapeutic Impact
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Assumpta Caixas, Principal Investigator, Corporacion Parc Tauli
Other Study IDs: 2025/5022
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Prader Willi Syndrome; Hyperphagia; Behavior Disorders
Keywords: Neuroimage; Artificial Intelligence; Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome; Hyperphagia; Mental Disorders | interventions — Human Growth Hormone; Eating

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Neuroimages of fMRI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patients with PWS: Adult (>18 y.o.) patients with genetically confirmed diagnosis of Prader-Willi syndrome.
  Interventions: Drug: GH treatment (Somatropin); Behavioral: Eating
- Healthy controls: Age and sex matched healthy controls
  Interventions: Behavioral: Eating
- Obese controls: Age and sex matched controls with obesity (BMI > 30)
  Interventions: Behavioral: Eating

INTERVENTIONS:
Drug: GH treatment (Somatropin) — Treatment with Somatropin (recombinant GH), with doses starting from 0.2 mg/day and adjusted as necessary.
  Groups: Patients with PWS
Behavioral: Eating — Allowing patients to break fasting.

SUMMARY:
The goal of this observational study is to explore brain network changes and identify patterns related to hyperphagia, hormonal treatment effects, and cognitive deficits in adults with Prader-Willi Syndrome (PWS). The main questions it aims to answer are:

* How are brain connectivity patterns altered in PWS patients compared to healthy and obese controls?
* How do brain network changes relate to hyperphagia and the response to growth hormone therapy?

Researchers will compare PWS patients to healthy and obese controls to see if there are significant differences in brain network connectivity before and after meals and growth hormone therapy. Ultimately, researchers will try to develop predictive models of treatment outcomes using AI and machine learning.

DETAILED DESCRIPTION:
Prader-Willi Syndrome (PWS) is a rare genetic condition marked by issues like constant hunger, obesity, hormonal imbalances, and cognitive difficulties. While studies have shown changes in brain connectivity in PWS patients, a complete understanding of these changes is still lacking. This project aims to explore brain network patterns in PWS using advanced AI techniques to better understand the impact of hyperphagia, hormonal treatments, and cognitive challenges.

This study will combine data from brain functional magnetic ressonance imaging (fMRI)), genetic data, hormonal levels, and clinical details; of 39 adults with PWS and 82 control participants (including 52 healthy and 30 obese controls). All participants are matched for age, sex, and BMI where applicable.

fMRI data has been obtained before and after meals, and/or before and after one year of growth hormone therapy.

Data quality will be assessed and summarize it using averages or percentages. Then, groups will be statistically compared to detect patterns related to hyperphagia and GH therapy.

Regarding Brain Connectivity, data from patients and controls will be compared, tracking how brain networks change after meals/GH therapy and applying advanced statistical methods to control errors.

Finally, using AI, models to predict treatment outcomes and brain network changes will be developed. These models will be tested and refined using different techniques to ensure reliability.

With this research, expected results are to identify unique brain patterns in PWS, uncover how these relate to symptoms like hyperphagia, and develop AI models to predict treatment outcomes. Ultimately, this research aims to improve our understanding of PWS and help develop better treatments.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed diagnosis of Prader-Willi Syndrome.
* Age older than 18 years old.

Exclusion Criteria:

* Age younger than 18 years old.
* Contraindications for fMRI.
* Visual defects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult (>18 y.o.) patients with PWS were selected from a cohort of patients who receive medical attention and follow-up at our hospital. Controls were also selected from hospital patients.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Functional connectivity patterns | Before and after the intervention (immediately after the end of the intervention for hunger, up to a year for GH).
  Brain connectivity patterns, particularly those related to hyperphagia and the response to growth hormone therapy in the case of PWS patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Consorci Corporació Sanitària Parc Taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No